CLINICAL TRIAL: NCT02905006
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose Ranging Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Study to Evaluate Safety and Efficacy of Different Doses of Bimekizumab in Patients With Chronic Plaque Psoriasis
Acronym: BE ABLE 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0010; 2016-001891-31 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis; Chronic Plaque Psoriasis; Bimekizumab
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Bimekizumab dosing regimen 1 (Experimental)
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab dosing regimen 2 (Experimental)
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab dosing regimen 3 (Experimental)
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab dosing regimen 4 (Experimental)
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab dosing regimen 5 (Experimental)
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will be randomized to receive a combination of injections of Bimekizumab.
  Other Names: UCB4940
  Arms: Bimekizumab dosing regimen 1; Bimekizumab dosing regimen 2; Bimekizumab dosing regimen 3; Bimekizumab dosing regimen 4; Bimekizumab dosing regimen 5
Other: Placebo — Subjects randomized to the placebo group, will receive a combination of several injections of Placebo to maintain the blinding.
  Arms: Bimekizumab dosing regimen 1; Bimekizumab dosing regimen 2; Bimekizumab dosing regimen 3; Bimekizumab dosing regimen 4; Placebo

SUMMARY:
This is a Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose ranging study to investigate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of Bimekizumab compared with placebo in adult subjects with moderate to severe chronic plaque psoriasis in order to guide the selection of doses and clinical indices in the Phase 3 development program.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Chronic plaque psoriasis for at least 6 months prior to Screening
* PASI (Psoriasis Area and Severity Index) >=12 and BSA (body surface area) >=10% and IGA (Investigator's Global Assessment) score 3 or greater on a 5-point scale
* Candidates for systemic psoriasis therapy and/or phototherapy and/or chemophototherapy
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception up till 20 weeks after last administration of study drug
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of study medication

Exclusion Criteria:

* Subjects with erythrodermic, guttate, pustular form of psoriasis, or drug-induced psoriasis
* Subject has any severe, progressive and/or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, gastrointestinal or neurological disease
* Subject has any significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol
* Subject taking prohibited psoriatic medications
* Subject receiving any live vaccines within 8 weeks prior to the Baseline and subjects receiving Bacillus Calmette-Guerin (BCG) vaccination within 1 year prior to study drug administration
* Subject has previously received treatment with any anti-interleukin-17 (anti-IL-17) therapy or has been exposed to more than 1 biological response modifier (limited to anti-tumor necrosis factor (TNF) or IL-12/23) for psoriatic arthritis or psoriasis prior to the Baseline
* Subject has any current sign or symptom that may indicate an active infection (except for common cold)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (41):
- United States (11):
  - Ps0010 711, Fremont, California
  - Ps0010 708, Los Angeles, California
  - Ps0010 706, Washington D.C., District of Columbia
  - Ps0010 704, West Des Moines, Iowa
  - Ps0010 718, Rochester, New York
  - Ps0010 738, Wilmington, North Carolina
  - Ps0010 736, Cleveland, Ohio
  - Ps0010 712, Portland, Oregon
  - Ps0010 733, Dallas, Texas
  - Ps0010 702, Houston, Texas
  - Ps0010 709, Houston, Texas
- Canada (8):
  - Ps0010 203, Surrey, British Columbia
  - Ps0010 204, Hamilton, Ontario
  - Ps0010 201, North Bay, Ontario
  - Ps0010 206, Peterborough, Ontario
  - Ps0010 205, Waterloo, Ontario
  - Ps0010 214, Québec, Quebec
  - Ps0010 209, Edmonton
  - Ps0010 214, Québec
- Czechia (4):
  - Ps0010 300, Ostrava Poruba
  - Ps0010 303, Pardubice
  - Ps0010 301, Prague
  - Ps0010 304, Prague
- Hungary (3):
  - Ps0010 404, Kecskemét
  - Ps0010 400, Orosháza
  - Ps0010 405, Szekszárd
- Japan (4):
  - Ps0010 502, Nagoya
  - Ps0010 501, Shinaga Wa-ku
  - Ps0010 503, Tokyo
  - Ps0010 504, Tokyo
- Poland (11):
  - Ps0010 600, Bialystok
  - Ps0010 611, Bialystok
  - Ps0010 605, Gdansk
  - Ps0010 610, Gdynia
  - Ps0010 604, Kielce
  - Ps0010 608, Krakow
  - Ps0010 606, Lublin
  - Ps0010 603, Podlaski
  - Ps0010 607, Warsaw
  - Ps0010 601, Wroclaw
  - Ps0010 609, Wroclaw

REFERENCES:
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2016 and concluded in July 2017.
Pre-assignment Details: The study included a 2-4 week Screening Period and a 12-week Treatment Period. Completed study was defined as completed the 12-week double-blind Treatment Period. After Treatment Period participants either enrolled in an extension study (PS0011) or entered a 20-week Safety Follow-Up Period.
  Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants randomized to the placebo group, received a combination of several injections of placebo, subcutaneously every 4 weeks (Q4W).
- Bimekizumab 64 mg Q4W: Participants were randomized to receive subcutaneous injections of 64 mg bimekizumab Q4W.
- Bimekizumab 160 mg Q4W: Participants were randomized to receive subcutaneous injections of 160 mg bimekizumab Q4W.
- Bimekizumab 160 mg w/ LD Q4W: Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W.
- Bimekizumab 320 mg Q4W: Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab Q4W.
- Bimekizumab 480 mg Q4W: Participants were randomized to receive subcutaneous injections of 480 mg bimekizumab Q4W.
Period: Overall Study
Arm/Group | Placebo | Bimekizumab 64 mg Q4W | Bimekizumab 160 mg Q4W | Bimekizumab 160 mg w/ LD Q4W | Bimekizumab 320 mg Q4W | Bimekizumab 480 mg Q4W
Started | 42 | 39 | 43 | 40 | 43 | 43
Completed Treatment Period | 37 | 36 | 38 | 34 | 40 | 39
Enrolled in Extension Study (PS0011) | 38 | 35 | 39 | 38 | 42 | 40
Entered Safety Follow-up Period | 4 | 4 | 4 | 2 | 1 | 3
Completed | 37 | 36 | 38 | 34 | 40 | 39
Not Completed | 5 | 3 | 5 | 6 | 3 | 4
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Screening exclusion criteria met | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lab withdrawal criterion met | 0 | 1 | 2 | 2 | 2 | 1
Not completed — Positive for Tuberculosis | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Subject positive for Hep B | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Patient moved abroad | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient randomized by mistake | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set, which consisted of all participants who received at least 1 dose of the study medication.
Arm/Group | Placebo | Bimekizumab 64 mg Q4W | Bimekizumab 160 mg Q4W | Bimekizumab 160 mg w/ LD Q4W | Bimekizumab 320 mg Q4W | Bimekizumab 480 mg Q4W | Total Title
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Between 18 and 65 years | 39 | 36 | 40 | 35 | 39 | 36 | 225
  >=65 years | 3 | 2 | 3 | 5 | 4 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.3) | 44.2 (13.8) | 43.4 (12.4) | 46.5 (15.2) | 42.6 (13.6) | 42.9 (15.2) | 44.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 11 | 11 | 15 | 14 | 87
  Male | 25 | 20 | 32 | 29 | 28 | 29 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Asian | 3 | 2 | 4 | 6 | 3 | 4 | 22
  Black | 0 | 1 | 0 | 1 | 1 | 0 | 3
  White | 39 | 35 | 39 | 33 | 39 | 38 | 223

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 90% or Higher Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received at least 1 dose of the study medication and had a valid measurement of the primary efficacy variable at Baseline.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (FAS): Participants randomized to the placebo group, received a combination of several injections of placebo, subcutaneously every 4 weeks (Q4W). Participants formed the Full Analysis Set (FAS).
- Bimekizumab 64 mg Q4W (FAS): Participants were randomized to receive subcutaneous injections of 64 mg bimekizumab Q4W. Participants formed the FAS.
- Bimekizumab 160 mg Q4W (FAS): Participants were randomized to receive subcutaneous injections of 160 mg bimekizumab Q4W. Participants formed the FAS.
- Bimekizumab 160 mg w/ LD Q4W (FAS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W. Participants formed the FAS.
- Bimekizumab 320 mg Q4W (FAS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab Q4W. Participants formed the FAS.
- Bimekizumab 480 mg Q4W (FAS): Participants were randomized to receive subcutaneous injections of 480 mg bimekizumab Q4W. Participants formed the FAS.
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 0 | 46.2 | 67.4 | 75.0 | 79.1 | 72.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic — P-value evaluating dose response excludes the BKZ Dose 3 group; is based on a logistic regression model with fixed effects for region, prior biologic exposure, continuous treatment variable with values of -2, -1, 0, 1, 2 for the remaining groups
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) (Clear or Almost Clear With at Least 2 Category Improvement From Baseline) Response at Week 12
Description: The Investigator's Global Assessment (IGA) measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 4.8 | 51.3 | 74.4 | 75.0 | 86.0 | 76.7
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); Test type: Superiority; p = 0.0001, Regression, Logistic; Confidence intervals, odds ratios, p-values derived from a logistic regression model with fixed effects for treatment, region, prior bio-exposure; Odds Ratio (OR) = 21.43, 95% CI 2-sided [4.51 to 101.88]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 63.21, 95% CI 2-sided [12.90 to 309.83]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 160 mg w/ LD Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 62.35, 95% CI 2-sided [12.61 to 308.29]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 130.35, 95% CI 2-sided [24.50 to 693.51]
Statistical Analysis 5: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 69.40, 95% CI 2-sided [14.07 to 342.40]

3. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) (Clear or Almost Clear With at Least 2 Category Improvement From Baseline) Response at Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 4.8 | 46.2 | 62.8 | 77.5 | 86.0 | 72.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); Test type: Superiority; p = 0.0003, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 18.23, 95% CI 2-sided [3.79 to 87.76]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 39.60, 95% CI 2-sided [8.19 to 191.59]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 160 mg w/ LD Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 77.27, 95% CI 2-sided [15.19 to 392.93]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 141.99, 95% CI 2-sided [26.26 to 767.72]
Statistical Analysis 5: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 58.52, 95% CI 2-sided [11.89 to 288.00]

4. Secondary Outcome: Percentage of Participants Achieving a 90% or Higher Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 0 | 41.0 | 58.1 | 67.5 | 86.0 | 69.8
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Fisher Exact — The placebo treatment group contained no PASI90 responders and as such the p-values for the pairwise comparisons are based upon the Fisher's exact test
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 160 mg w/ LD Q4W (FAS); Test type: Superiority; p < 0.0001, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Fisher Exact — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Fisher Exact — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving a 75% or Higher Improvement in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline. This is a scoring system that averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale), and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 4.8 | 61.5 | 81.4 | 85.0 | 93.0 | 83.7
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 32.65, 95% CI 2-sided [6.82 to 156.38]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 94.51, 95% CI 2-sided [18.54 to 481.86]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 160 mg w/ LD Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 117.66, 95% CI 2-sided [22.08 to 626.89]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 280.76, 95% CI 2-sided [44.06 to 1789.24]
Statistical Analysis 5: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 107.83, 95% CI 2-sided [20.82 to 558.57]

6. Secondary Outcome: Percentage of Participants Achieving a 100% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72. The PASI 100 response rate at Week 12 is measured as the percentage of participants who achieved 100% improvement from baseline PASI at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Bimekizumab 64 mg Q4W (FAS) | Bimekizumab 160 mg Q4W (FAS) | Bimekizumab 160 mg w/ LD Q4W (FAS) | Bimekizumab 320 mg Q4W (FAS) | Bimekizumab 480 mg Q4W (FAS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 0 | 28.2 | 27.9 | 60.0 | 55.8 | 48.8
Statistical Analysis 1: Comparison: Placebo (FAS) vs Bimekizumab 64 mg Q4W (FAS); The placebo treatment group contained no PASI100 responders and as such the p-values for the pairwise comparisons are based upon the Fisher's exact test; Test type: Superiority; p = 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo (FAS) vs Bimekizumab 160 mg Q4W (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0002, Fisher Exact
Statistical Analysis 3: Comparison: Placebo (FAS) vs Bimekizumab 160 mg w/ LD Q4W (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 4: Comparison: Placebo (FAS) vs Bimekizumab 320 mg Q4W (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 5: Comparison: Placebo (FAS) vs Bimekizumab 480 mg Q4W (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Fisher Exact

7. Secondary Outcome: Plasma Concentrations of Bimekizumab During the Study
Description: Bimekizumab plasma concentration was expressed in micrograms per milliliter (μg/mL).
  Values Below Limit of Quantification (BLQ) were replaced by the value of lower limit of quantification (LLOQ) divided by 2 = 0.075 μg/mL in the calculations of geometric mean and confidence intervals (CIs). Geometric mean was only calculated if at least two-thirds of the concentrations were quantified at the respective time point.
Time Frame: Baseline (Week 0), Week 1, Week 2, Week 4, Week 8, Week 12, and Safety Follow-Up visit (20 weeks after the last dose)
Population: The Pharmacokinetics Per-Protocol Set (PK-PPS) consisted of all randomized participants who took at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration postdose and had no important protocol deviations affecting the PK variables.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Bimekizumab 64 mg Q4W (PK-PPS): Participants were randomized to receive subcutaneous injections of 64 mg bimekizumab Q4W. Participants formed the PK-PPS.
- Bimekizumab 160 mg Q4W (PK-PPS): Participants were randomized to receive subcutaneous injections of 160 mg bimekizumab Q4W. Participants formed the PK-PPS.
- Bimekizumab 160 mg w/ LD Q4W (PK-PPS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W. Participants formed the PK-PPS.
- Bimekizumab 320 mg Q4W (PK-PPS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab Q4W. Participants formed the PK-PPS.
- Bimekizumab 480 mg Q4W (PK-PPS): Participants were randomized to receive subcutaneous injections of 480 mg bimekizumab Q4W. Participants formed the PK-PPS.
Arm/Group | Bimekizumab 64 mg Q4W (PK-PPS) | Bimekizumab 160 mg Q4W (PK-PPS) | Bimekizumab 160 mg w/ LD Q4W (PK-PPS) | Bimekizumab 320 mg Q4W (PK-PPS) | Bimekizumab 480 mg Q4W (PK-PPS)
Number analyzed (Participants) | 39 | 42 | 40 | 43 | 43
µg/mL
  Baseline | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment. | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment. | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment. | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment. | NA [NA to NA] — Values were below the level of detection; Participants had no prior BKZ treatment.
  Week 1 | 4.4490 [3.7526 to 5.2746] | 9.2481 [6.9779 to 12.2569] | 20.7892 [14.9192 to 28.9688] | 21.8622 [16.0624 to 29.7563] | 31.8019 [23.3488 to 43.3154]
  Week 2: number analyzed (Participants) | 39 | 41 | 39 | 42 | 42
  Week 2 | 3.4704 [3.0167 to 3.9923] | 8.6862 [7.5316 to 10.0179] | 19.0428 [16.5381 to 21.9267] | 19.0324 [16.8925 to 21.4434] | 27.5641 [23.8485 to 31.8586]
  Week 4: number analyzed (Participants) | 39 | 41 | 39 | 41 | 40
  Week 4 | 2.1282 [1.8398 to 2.4617] | 5.3751 [4.5233 to 6.3872] | 11.2903 [9.4809 to 13.4450] | 11.9194 [10.4503 to 13.5951] | 17.1811 [14.7612 to 19.9977]
  Week 8: number analyzed (Participants) | 38 | 38 | 37 | 40 | 40
  Week 8 | 2.3069 [1.7780 to 2.9931] | 7.1859 [5.3747 to 9.6075] | 10.2208 [8.8561 to 11.7957] | 16.3187 [13.9947 to 19.0285] | 23.3285 [19.8863 to 27.3665]
  Week 12: number analyzed (Participants) | 38 | 38 | 33 | 40 | 39
  Week 12 | 2.3121 [1.6037 to 3.3335] | 9.5278 [8.0614 to 11.2608] | 10.2557 [8.6807 to 12.1165] | 18.3166 [15.1652 to 22.1228] | 28.0908 [23.2463 to 33.9448]
  SFU: number analyzed (Participants) | 4 | 4 | 2 | 1 | 3
  SFU | NA [NA to NA] — Values were below the level of detection. | NA [NA to NA] — Values were below the level of detection. | NA [NA to NA] — Values were below the level of detection. | NA [NA to NA] — Values were below the level of detection. | 0.5165 [0.0032 to 84.5222]

8. Secondary Outcome: Population PK (Apparent Total Clearance (CL/F)) of Bimekizumab
Description: The data were presented as population estimates of CL/F. Given the sparse nature of PK sampling, CL/F cannot be estimated for each treatment group.
  It was prespecified in the data analysis plan to combine doses to perform Population PK and PK/PD analysis based on a prior determination that the PK parameters are not dose-dependent.
Time Frame: From Baseline (Week 0) until Safety Follow-Up Visit (20 weeks after the last dose; Up to Week 28)
Population: The PK-PPS consisted of all randomized participants who took at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration postdose and had no important protocol deviations affecting the PK variables. Given the sparse nature of PK sampling, CL/F cannot be estimated for each treatment group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/Day
Groups:
- All Participants (PK-PPS): Participants were randomized to receive subcutaneous injections of placebo or bimekizumab in different dosages: 64 mg Q4W, 160 mg Q4W, 320 mg loading dose at Baseline followed by 160 mg Q4W, 320 mg Q4W, 480 mg Q4W during the 12-week Treatment Period. Participants formed the PK-PPS.
Arm/Group | All Participants (PK-PPS)
Number analyzed (Participants) | 249
L/Day | 0.362 (41.7)

9. Secondary Outcome: Population PK (Apparent Volume of Distribution (V/F)) of Bimekizumab
Description: The data were presented as population estimates of V/F. Given the sparse nature of PK sampling, V/F cannot be estimated for each treatment group.
  It was prespecified in the data analysis plan to combine doses to perform Population PK and PK/PD analysis based on a prior determination that the PK parameters are not dose-dependent.
Time Frame: From Baseline (Week 0) until Safety Follow-Up Visit (20 weeks after the last dose; Up to Week 28)
Population: The PK-PPS consisted of all randomized participants who took at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration postdose and had no important protocol deviations affecting the PK variables. Given the sparse nature of PK sampling, V/F cannot be estimated for each treatment group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | All Participants (PK-PPS)
Number analyzed (Participants) | 249
liters | 11.5 (146)

10. Secondary Outcome: Concentration of Bimekizumab Leading to 50% of Maximum Effect (EC50)
Description: The data were presented as population estimates of EC50. EC50 was estimated based on all available data and cannot be derived for each treatment arm.
  It was prespecified in the data analysis plan to combine doses to perform Population PK and PK/PD analysis based on a prior determination that the PK parameters are not dose-dependent.
Time Frame: From Baseline (Week 0) until Safety Follow-Up Visit (20 weeks after the last dose; Up to Week 28)
Population: The PK-PPS consisted of all randomized participants who took at least 1 dose of the IMP and provided at least 1 quantifiable plasma concentration postdose and had no important protocol deviations affecting the PK variables. EC50 was estimated based on all available data and cannot be derived for each treatment arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | All Participants (PK-PPS)
Number analyzed (Participants) | 249
µg/mL | 0.55 (126)

11. Secondary Outcome: Percentage of Participants With a Positive Anti-bimekizumab Antibody (AbAb) Status Prior to Study Treatment
Description: Antibody positive status prior study treatment was defined as having an antibody level greater than (>) 28.5% at Baseline (Week 0).
Time Frame: Baseline (Week 0)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- Placebo (PK-PPS): Participants randomized to the placebo group, received a combination of several injections of placebo, subcutaneously every 4 weeks (Q4W). Participants formed the Pharmacokinetics Per-Protocol Set (PK-PPS).
Arm/Group | Placebo (PK-PPS) | Bimekizumab 64 mg Q4W (PK-PPS) | Bimekizumab 160 mg Q4W (PK-PPS) | Bimekizumab 160 mg w/ LD Q4W (PK-PPS) | Bimekizumab 320 mg Q4W (PK-PPS) | Bimekizumab 480 mg Q4W (PK-PPS)
Number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
percentage of participants | 0 | 0 | 0 | 2.5 | 0 | 0

12. Secondary Outcome: Percentage of Participants With an Overall Positive Anti-bimekizumab Antibody (AbAb) Status Following Study Treatment
Description: Overall antibody positive was defined as having a value of > 28.5% at any time in the Treatment Period. The Treatment Period did not include Baseline/pretreatment samples.
Time Frame: From Week 4 until the Safety Follow-Up visit (20 weeks after the last dose; Up to Week 28)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (PK-PPS) | Bimekizumab 64 mg Q4W (PK-PPS) | Bimekizumab 160 mg Q4W (PK-PPS) | Bimekizumab 160 mg w/ LD Q4W (PK-PPS) | Bimekizumab 320 mg Q4W (PK-PPS) | Bimekizumab 480 mg Q4W (PK-PPS)
Number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
percentage of participants | 0 | 10.3 | 4.8 | 5.0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Study
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IMP.
Time Frame: From Screening to End of Safety Follow-up (up to Week 32)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Participants randomized to the placebo group, received a combination of several injections of placebo, subcutaneously every 4 weeks (Q4W). Participants formed the Safety Set (SS).
- Bimekizumab 64 mg Q4W (SS): Participants were randomized to receive subcutaneous injections of 64 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 160 mg Q4W (SS): Participants were randomized to receive subcutaneous injections of 160 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 160 mg w/ LD Q4W (SS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 320 mg Q4W (SS): Participants were randomized to receive subcutaneous injections of 320 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 480 mg Q4W (SS): Participants were randomized to receive subcutaneous injections of 480 mg bimekizumab Q4W. Participants formed the SS.
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 38.1 | 76.9 | 55.8 | 65.0 | 60.5 | 60.5

14. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Study by Severity
Description: as for outcome 13
Time Frame: From Screening to End of Safety Follow-up (up to Week 32)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants
  Mild | 11.9 | 43.6 | 27.9 | 22.5 | 39.5 | 44.2
  Moderate | 26.2 | 30.8 | 27.9 | 40.0 | 20.9 | 11.6
  Severe | 0 | 2.6 | 0 | 2.5 | 0 | 4.7

15. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Platelets)
Description: Platelets was measured in number of platelets per liter (10^9/L).
Time Frame: Baseline (Week 0), Week 1, Week 2, Week 4, Week 6, Week 8, Week 12, and Safety Follow-Up visit (20 weeks after the last dose)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
10^9 platelets per liter
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Week 1 | 12.1 (34.7) | 3.2 (21.0) | -4.6 (30.8) | -14.0 (30.8) | 3.5 (25.2) | -0.1 (35.0)
  Week 2: number analyzed (Participants) | 41 | 39 | 40 | 39 | 41 | 41
  Week 2 | 6.4 (37.8) | -8.6 (26.8) | -5.6 (36.4) | -8.9 (27.8) | 7.8 (31.2) | -3.9 (41.8)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 40 | 40
  Week 4 | -0.1 (32.0) | -5.8 (28.3) | -8.6 (40.1) | -11.4 (21.8) | -7.0 (28.9) | -7.5 (36.8)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 39 | 40
  Week 6 | 5.6 (47.5) | -5.2 (26.3) | -13.6 (34.3) | -5.6 (30.3) | -0.3 (44.0) | -7.6 (37.3)
  Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Week 8 | 6.9 (37.6) | -2.3 (44.7) | -6.1 (43.7) | 6.3 (35.6) | 0.7 (39.5) | -4.7 (36.4)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Week 12 | 2.8 (36.7) | -6.0 (36.2) | -13.2 (40.1) | -3.6 (37.5) | -5.4 (36.1) | -5.5 (38.8)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 14.8 (33.3) | -30.3 (71.6) | 7.8 (20.0) | -33.0 (31.1) | 39.0 (NA) — Value was not evaluable because only one participant was analyzed. | 39.3 (27.4)

16. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration, Hemoglobin)
Description: Erythrocytes mean corpuscular hemoglobin (HGB) concentration and hemoglobin were measured in grams per liter (g/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
g/L
  Ery. mean corpuscular HGB Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Ery. mean corpuscular HGB Week 1 | 0.1 (8.1) | -2.0 (10.3) | -0.3 (8.8) | -1.0 (11.6) | 0.5 (8.6) | 0.3 (8.1)
  Ery. mean corpuscular HGB Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Ery. mean corpuscular HGB Week 2 | 0.1 (7.9) | 1.1 (6.6) | 1.6 (9.4) | -0.3 (9.8) | 2.6 (7.9) | 1.8 (8.8)
  Ery. mean corpuscular HGB Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Ery. mean corpuscular HGB Week 4 | -0.2 (9.1) | 0.2 (8.3) | -0.1 (9.9) | -2.9 (6.3) | 0.1 (8.0) | -0.4 (11.7)
  Ery. mean corpuscular HGB Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Ery. mean corpuscular HGB Week 6 | -2.5 (11.0) | -1.7 (8.6) | -0.5 (9.4) | -2.9 (7.0) | -0.5 (7.8) | -1.3 (8.9)
  Ery. mean corpuscular HGB Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Ery. mean corpuscular HGB Week 8 | -2.2 (8.0) | -1.4 (12.7) | 0.3 (10.3) | -2.5 (7.9) | -2.1 (9.2) | -2.9 (9.2)
  Ery. mean corpuscular HGB Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Ery. mean corpuscular HGB Week 12 | -6.3 (12.5) | -2.2 (14.7) | -1.6 (9.1) | -4.5 (10.1) | -2.0 (12.7) | -3.6 (13.7)
  Ery. mean corpuscular HGB SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Ery. mean corpuscular HGB SFU | -12.5 (11.0) | 5.3 (26.2) | -5.5 (10.6) | -9.5 (7.8) | -2.0 (NA) — Value was not evaluable because only one participant was analyzed. | -22.0 (18.0)
  Hemoglobin Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Hemoglobin Week 1 | -2.9 (7.3) | 0.1 (6.1) | 1.0 (6.8) | -2.6 (5.2) | -1.0 (7.0) | -0.8 (5.0)
  Hemoglobin Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Hemoglobin Week 2 | -3.0 (6.7) | 0.5 (5.3) | 0.6 (6.0) | -1.5 (7.5) | -1.1 (7.0) | 0.5 (6.6)
  Hemoglobin Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Hemoglobin Week 4 | -2.9 (8.2) | 0.8 (6.1) | -0.9 (6.2) | -2.1 (5.9) | -1.8 (8.7) | -0.4 (6.3)
  Hemoglobin Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Hemoglobin Week 6 | -2.4 (7.8) | 0.7 (6.3) | -0.3 (6.6) | -1.2 (4.8) | -2.1 (8.4) | 0.9 (6.3)
  Hemoglobin Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Hemoglobin Week 8 | -2.7 (8.0) | 1.1 (7.6) | 0.8 (7.1) | -0.6 (7.5) | -1.8 (8.1) | 0.9 (6.5)
  Hemoglobin Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Hemoglobin Week 12 | -1.8 (9.1) | 3.2 (9.6) | -0.1 (8.1) | -1.0 (8.5) | -1.2 (9.3) | 0.3 (7.1)
  Hemoglobin SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Hemoglobin SFU | -4.8 (7.4) | 7.8 (31.0) | -6.5 (4.7) | -8.5 (2.1) | 6.0 (NA) — Value was not evaluable because only one participant was analyzed. | -6.7 (11.0)

17. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes Mean Corpuscular Hemoglobin (HGB))
Description: Erythrocytes mean corpuscular hemoglobin (HGB) was measured in picograms (pg).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
picograms (pg)
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Week 1 | -0.09 (0.57) | -0.01 (0.56) | -0.10 (0.55) | 0.07 (0.51) | -0.09 (0.87) | 0.00 (0.53)
  Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Week 2 | -0.04 (0.59) | 0.04 (0.54) | 0.05 (0.49) | 0.10 (0.78) | -0.03 (0.60) | 0.14 (0.54)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Week 4 | -0.07 (0.66) | 0.10 (0.84) | -0.07 (0.63) | -0.01 (0.42) | -0.10 (0.68) | 0.04 (0.50)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | -0.17 (0.64) | -0.09 (0.84) | -0.16 (0.61) | -0.11 (0.47) | -0.12 (0.84) | -0.04 (0.60)
  Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Week 8 | -0.19 (0.64) | 0.09 (1.09) | -0.16 (1.10) | -0.16 (0.64) | -0.26 (0.99) | -0.16 (0.53)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Week 12 | -0.34 (0.71) | 0.09 (1.53) | -0.08 (0.58) | -0.14 (0.66) | -0.09 (1.14) | -0.16 (0.67)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | -0.33 (0.79) | 2.93 (6.66) | -0.15 (0.17) | -0.55 (0.78) | 0.70 (NA) — Value was not evaluable because only one participant was analyzed. | -0.60 (1.10)

18. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes Mean Corpuscular Volume)
Description: Erythrocytes mean corpuscular volume was measured in femtolitres (fL).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: femtolitres (fL)
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
femtolitres (fL)
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Week 1 | -0.35 (1.55) | 0.52 (2.29) | -0.25 (1.64) | 0.51 (2.63) | -0.23 (2.14) | -0.04 (1.37)
  Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Week 2 | -0.14 (1.65) | -0.16 (1.31) | -0.33 (1.96) | 0.31 (1.32) | -0.64 (1.40) | -0.05 (1.60)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Week 4 | -0.11 (1.60) | 0.23 (1.89) | -0.25 (1.81) | 0.67 (1.76) | -0.10 (1.64) | 0.22 (2.87)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | 0.20 (2.84) | 0.14 (2.47) | -0.29 (1.90) | 0.39 (1.79) | -0.02 (1.92) | 0.25 (1.85)
  Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Week 8 | 0.05 (2.11) | 0.71 (2.88) | -0.54 (2.57) | 0.16 (2.57) | -0.02 (2.29) | 0.36 (2.37)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Week 12 | 0.76 (3.81) | 0.87 (3.23) | 0.17 (2.39) | 0.78 (2.55) | 0.47 (2.88) | 0.51 (3.89)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 2.58 (5.10) | 7.80 (14.07) | 0.90 (2.38) | 0.85 (0.35) | 2.80 (NA) — Value was not evaluable because only one participant was analyzed. | 4.87 (8.46)

19. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Erythrocytes)
Description: Erythrocytes was measured in number of red blood cells per liter (10^12/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: 10^12 red blood cells per liter
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
10^12 red blood cells per liter
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Week 1 | -0.081 (0.282) | 0.004 (0.213) | 0.047 (0.238) | -0.095 (0.184) | -0.029 (0.259) | -0.026 (0.178)
  Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Week 2 | -0.088 (0.220) | 0.010 (0.193) | 0.014 (0.215) | -0.060 (0.282) | -0.041 (0.231) | -0.001 (0.232)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Week 4 | -0.085 (0.274) | 0.019 (0.217) | -0.018 (0.193) | -0.066 (0.215) | -0.053 (0.281) | -0.015 (0.216)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | -0.053 (0.277) | 0.038 (0.218) | 0.011 (0.243) | -0.019 (0.145) | -0.060 (0.278) | 0.035 (0.224)
  Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Week 8 | -0.062 (0.320) | 0.022 (0.245) | 0.048 (0.219) | 0.009 (0.224) | -0.028 (0.240) | 0.056 (0.238)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Week 12 | -0.007 (0.314) | 0.092 (0.258) | 0.011 (0.271) | -0.005 (0.297) | -0.036 (0.297) | 0.039 (0.228)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | -0.090 (0.346) | -0.135 (0.184) | -0.195 (0.165) | -0.215 (0.035) | 0.080 (NA) — Value was not evaluable because only one participant was analyzed. | -0.123 (0.491)

20. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Hematocrit)
Description: Hematocrit was measured in volume percentage (%) of red blood cells in blood.
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: volume % of red blood cells
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
volume % of red blood cells
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Week 1 | -0.88 (2.49) | 0.27 (2.07) | 0.33 (2.31) | -0.58 (2.14) | -0.36 (2.31) | -0.23 (1.62)
  Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Week 2 | -0.86 (2.02) | 0.00 (1.65) | -0.04 (2.15) | -0.42 (2.61) | -0.65 (2.09) | -0.02 (2.03)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Week 4 | -0.81 (2.40) | 0.24 (2.07) | -0.26 (1.86) | -0.26 (1.80) | -0.48 (2.57) | -0.03 (2.02)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | -0.33 (2.46) | 0.41 (1.88) | -0.04 (2.18) | 0.02 (1.73) | -0.51 (2.59) | 0.44 (1.90)
  Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Week 8 | -0.52 (2.37) | 0.55 (2.51) | 0.18 (1.84) | 0.14 (2.61) | -0.22 (2.46) | 0.67 (2.03)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 35 | 40 | 38
  Week 12 | 0.32 (2.87) | 1.25 (2.29) | 0.18 (2.57) | 0.30 (2.99) | -0.05 (2.75) | 0.59 (2.02)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 0.20 (1.44) | 1.98 (6.92) | -1.20 (1.90) | -1.50 (0.14) | 2.10 (NA) — Value was not evaluable because only one participant was analyzed. | 1.00 (0.85)

21. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Hematology Parameters (Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils)
Description: Basophils, eosinophils, leukocytes, lymphocytes, monocytes and neutrophils were measured in number of white blood cells per liter (10^9/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: 10^9 white blood cells per liter
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
10^9 white blood cells per liter
  Basophils Week 1: number analyzed (Participants) | 42 | 39 | 41 | 40 | 43 | 42
  Basophils Week 1 | 0.01 (0.03) | 0.01 (0.03) | 0.00 (0.03) | 0.01 (0.03) | 0.00 (0.04) | 0.01 (0.03)
  Basophils Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Basophils Week 2 | 0.00 (0.02) | 0.00 (0.04) | 0.01 (0.04) | 0.01 (0.04) | 0.01 (0.04) | 0.00 (0.03)
  Basophils Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Basophils Week 4 | 0.00 (0.03) | 0.00 (0.05) | 0.00 (0.03) | 0.01 (0.02) | 0.01 (0.05) | 0.00 (0.04)
  Basophils Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Basophils Week 6 | 0.01 (0.03) | 0.00 (0.04) | 0.00 (0.04) | 0.01 (0.02) | 0.00 (0.04) | 0.00 (0.04)
  Basophils Week 8: number analyzed (Participants) | 39 | 37 | 37 | 34 | 40 | 40
  Basophils Week 8 | 0.00 (0.04) | -0.01 (0.04) | 0.02 (0.01) | 0.00 (0.00) | 0.02 (0.04) | 0.00 (0.05)
  Basophils Week 12: number analyzed (Participants) | 38 | 38 | 37 | 34 | 40 | 38
  Basophils Week 12 | 0.00 (0.03) | 0.00 (0.04) | 0.01 (0.03) | 0.00 (0.02) | 0.01 (0.04) | 0.00 (0.04)
  Basophils SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Basophils SFU | 0.03 (0.05) | -0.03 (0.05) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (NA) — Value was not evaluable because only one participant was analyzed. | 0.03 (0.06)
  Eosinophils Week 1: number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 42
  Eosinophils Week 1 | 0.02 (0.06) | 0.02 (0.12) | 0.01 (0.07) | 0.04 (0.10) | 0.02 (0.11) | -0.02 (0.12)
  Eosinophils Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Eosinophils Week 2 | 0.02 (0.08) | 0.04 (0.26) | 0.00 (0.08) | 0.05 (0.11) | 0.00 (0.11) | 0.01 (0.11)
  Eosinophils Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Eosinophils Week 4 | 0.03 (0.09) | 0.04 (0.26) | 0.01 (0.08) | 0.02 (0.11) | 0.03 (0.09) | 0.00 (0.18)
  Eosinophils Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Eosinophils Week 6 | 0.04 (0.10) | 0.02 (0.19) | 0.00 (0.08) | 0.01 (0.09) | 0.05 (0.16) | -0.01 (0.17)
  Eosinophils Week 8: number analyzed (Participants) | 39 | 37 | 37 | 34 | 40 | 40
  Eosinophils Week 8 | 0.01 (0.09) | 0.01 (0.18) | 0.01 (0.08) | 0.04 (0.17) | 0.05 (0.18) | -0.03 (0.16)
  Eosinophils Week 12: number analyzed (Participants) | 38 | 38 | 37 | 34 | 40 | 38
  Eosinophils Week 12 | 0.02 (0.09) | 0.03 (0.22) | 0.00 (0.09) | 0.00 (0.08) | 0.03 (0.13) | -0.03 (0.11)
  Eosinophils SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Eosinophils SFU | 0.05 (0.06) | 0.08 (0.10) | 0.10 (0.00) | 0.00 (0.00) | -0.10 (NA) — Value was not evaluable because only one participant was analyzed. | 0.07 (0.06)
  Leukocytes Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Leukocytes Week 1 | 0.16 (1.30) | -0.59 (1.34) | -0.15 (1.43) | -0.63 (1.82) | -0.19 (1.51) | -0.48 (0.90)
  Leukocytes Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Leukocytes Week 2 | 0.18 (1.36) | -0.56 (1.31) | -0.22 (1.43) | -0.42 (1.34) | -0.31 (1.80) | -0.46 (1.29)
  Leukocytes Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Leukocytes Week 4 | 0.17 (1.51) | -0.36 (1.31) | -0.23 (1.38) | -0.54 (1.14) | -0.36 (1.73) | -0.34 (1.24)
  Leukocytes Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Leukocytes Week 6 | -0.22 (1.25) | -0.50 (1.95) | -0.47 (1.49) | -0.57 (1.34) | -0.45 (2.02) | -0.45 (1.12)
  Leukocytes Week 8: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 40
  Leukocytes Week 8 | -0.10 (1.34) | -0.67 (1.55) | -0.24 (1.94) | -0.37 (1.55) | -0.30 (1.76) | -0.45 (0.87)
  Leukocytes Week 12: number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 38
  Leukocytes Week 12 | 0.00 (1.37) | -0.28 (1.68) | -0.47 (1.67) | -0.51 (1.41) | -0.50 (1.44) | -0.48 (1.09)
  Leukocytes SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Leukocytes SFU | -0.05 (0.98) | 1.15 (2.54) | 0.95 (1.43) | -0.65 (0.78) | 0.20 (NA) — Value was not evaluable because only one participant was analyzed. | 0.30 (0.40)
  Lymphocytes Week 1: number analyzed (Participants) | 42 | 39 | 41 | 40 | 43 | 42
  Lymphocytes Week 1 | 0.12 (0.36) | -0.05 (0.30) | 0.15 (0.42) | 0.13 (0.34) | 0.14 (0.46) | 0.00 (0.45)
  Lymphocytes Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Lymphocytes Week 2 | 0.08 (0.32) | -0.11 (0.30) | 0.09 (0.34) | 0.09 (0.40) | 0.12 (0.34) | -0.08 (0.37)
  Lymphocytes Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Lymphocytes Week 4 | 0.06 (0.40) | -0.04 (0.33) | 0.15 (0.43) | 0.08 (0.42) | 0.11 (0.36) | 0.06 (0.36)
  Lymphocytes Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Lymphocytes Week 6 | 0.08 (0.46) | -0.08 (0.43) | 0.03 (0.31) | 0.04 (0.43) | 0.05 (0.37) | -0.05 (0.40)
  Lymphocytes Week 8: number analyzed (Participants) | 39 | 37 | 37 | 34 | 40 | 40
  Lymphocytes Week 8 | 0.02 (0.37) | -0.04 (0.31) | 0.09 (0.40) | 0.11 (0.33) | 0.15 (0.45) | 0.06 (0.42)
  Lymphocytes Week 12: number analyzed (Participants) | 38 | 38 | 37 | 34 | 40 | 38
  Lymphocytes Week 12 | 0.08 (0.38) | 0.01 (0.35) | 0.06 (0.38) | 0.07 (0.48) | 0.14 (0.38) | -0.04 (0.37)
  Lymphocytes SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Lymphocytes SFU | 0.25 (0.24) | 0.25 (0.40) | 0.23 (0.19) | 0.25 (0.21) | 0.00 (NA) — Value was not evaluable because only one participant was analyzed. | 0.50 (0.44)
  Monocytes Week 1: number analyzed (Participants) | 42 | 39 | 41 | 40 | 43 | 42
  Monocytes Week 1 | 0.02 (0.16) | -0.01 (0.12) | 0.02 (0.15) | 0.02 (0.11) | 0.02 (0.17) | -0.03 (0.14)
  Monocytes Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Monocytes Week 2 | 0.00 (0.14) | -0.04 (0.13) | 0.00 (0.14) | 0.04 (0.15) | -0.04 (0.17) | -0.03 (0.15)
  Monocytes Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Monocytes Week 4 | 0.03 (0.16) | -0.01 (0.11) | 0.01 (0.15) | 0.03 (0.13) | -0.01 (0.17) | 0.02 (0.17)
  Monocytes Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Monocytes Week 6 | 0.01 (0.15) | -0.01 (0.18) | 0.02 (0.15) | 0.00 (0.11) | -0.02 (0.22) | -0.03 (0.18)
  Monocytes Week 8: number analyzed (Participants) | 39 | 37 | 37 | 34 | 40 | 40
  Monocytes Week 8 | -0.02 (0.15) | -0.03 (0.11) | 0.00 (0.16) | -0.01 (0.14) | -0.04 (0.17) | -0.02 (0.15)
  Monocytes Week 12: number analyzed (Participants) | 38 | 38 | 37 | 34 | 40 | 38
  Monocytes Week 12 | 0.01 (0.16) | 0.00 (0.14) | -0.02 (0.15) | -0.01 (0.18) | -0.07 (0.17) | -0.01 (0.14)
  Monocytes SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Monocytes SFU | 0.10 (0.22) | 0.10 (0.22) | 0.03 (0.10) | 0.00 (0.00) | -0.30 (NA) — Value was not evaluable because only one participant was analyzed. | -0.07 (0.21)
  Neutrophils Week 1: number analyzed (Participants) | 42 | 39 | 41 | 40 | 43 | 42
  Neutrophils Week 1 | -0.02 (1.16) | -0.55 (1.12) | -0.32 (1.25) | -0.81 (1.81) | -0.37 (1.20) | -0.44 (0.76)
  Neutrophils Week 2: number analyzed (Participants) | 41 | 38 | 41 | 39 | 40 | 41
  Neutrophils Week 2 | 0.09 (1.29) | -0.43 (1.05) | -0.31 (1.33) | -0.59 (1.09) | -0.41 (1.64) | -0.36 (1.13)
  Neutrophils Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Neutrophils Week 4 | 0.04 (1.30) | -0.35 (1.07) | -0.39 (1.31) | -0.68 (1.02) | -0.48 (1.60) | -0.40 (1.18)
  Neutrophils Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Neutrophils Week 6 | -0.36 (0.98) | -0.43 (1.64) | -0.49 (1.38) | -0.54 (1.16) | -0.50 (1.78) | -0.36 (1.01)
  Neutrophils Week 8: number analyzed (Participants) | 39 | 37 | 37 | 34 | 40 | 40
  Neutrophils Week 8 | -0.13 (1.18) | -0.61 (1.40) | -0.34 (1.72) | -0.57 (1.28) | -0.45 (1.61) | -0.47 (0.80)
  Neutrophils Week 12: number analyzed (Participants) | 38 | 38 | 37 | 34 | 40 | 38
  Neutrophils Week 12 | -0.11 (1.17) | -0.33 (1.50) | -0.49 (1.50) | -0.57 (1.20) | -0.59 (1.28) | -0.39 (0.93)
  Neutrophils SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Neutrophils SFU | -0.45 (0.79) | 0.75 (1.88) | 0.65 (1.20) | -0.95 (0.49) | 0.50 (NA) — Value was not evaluable because only one participant was analyzed. | -0.13 (0.38)

22. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Calcium, Chloride, Potassium, Magnesium, Sodium, Urea Nitrogen, Cholesterol, Glucose)
Description: Calcium, chloride, potassium, magnesium, sodium, urea nitrogen, cholesterol and glucose were measured in millimoles per liter (mmol/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
mmol/L
  Calcium Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Calcium Week 1 | -0.010 (0.076) | 0.011 (0.088) | -0.021 (0.126) | -0.017 (0.076) | 0.000 (0.077) | -0.010 (0.080)
  Calcium Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Calcium Week 2 | -0.003 (0.082) | 0.034 (0.094) | -0.007 (0.092) | 0.004 (0.074) | 0.006 (0.088) | -0.006 (0.085)
  Calcium Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Calcium Week 4 | -0.029 (0.073) | 0.012 (0.099) | -0.020 (0.106) | -0.008 (0.074) | 0.005 (0.099) | -0.010 (0.084)
  Calcium Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Calcium Week 6 | -0.033 (0.070) | 0.009 (0.079) | -0.019 (0.091) | -0.008 (0.092) | -0.026 (0.086) | -0.027 (0.100)
  Calcium Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Calcium Week 8 | -0.023 (0.084) | 0.001 (0.106) | -0.027 (0.099) | 0.019 (0.089) | -0.002 (0.089) | -0.016 (0.084)
  Calcium Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Calcium Week 12 | -0.011 (0.095) | 0.025 (0.092) | -0.038 (0.120) | 0.001 (0.093) | -0.019 (0.121) | -0.001 (0.092)
  Calcium SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Calcium SFU | -0.095 (0.083) | -0.050 (0.109) | -0.073 (0.045) | -0.125 (0.134) | 0.020 (NA) — Value was not evaluable because only one participant was analyzed. | 0.020 (0.193)
  Chloride Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Chloride Week 1 | 0.5 (1.8) | 0.6 (2.0) | 0.6 (2.3) | 0.6 (2.5) | 0.3 (2.1) | 0.1 (1.8)
  Chloride Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Chloride Week 2 | 0.0 (2.3) | 0.1 (2.4) | -0.3 (2.2) | 0.4 (2.3) | 0.5 (2.1) | 0.1 (1.9)
  Chloride Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Chloride Week 4 | 0.1 (1.8) | 0.8 (2.1) | 0.0 (2.5) | 0.2 (2.3) | -0.1 (2.6) | -0.1 (1.9)
  Chloride Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Chloride Week 6 | -0.1 (2.1) | 0.0 (2.3) | -0.6 (1.7) | 0.0 (2.4) | -0.1 (3.0) | 0.1 (2.0)
  Chloride Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Chloride Week 8 | 0.2 (2.1) | 0.3 (2.3) | 0.3 (2.0) | -0.1 (2.9) | 0.1 (2.4) | 0.1 (2.3)
  Chloride Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Chloride Week 12 | 0.3 (1.7) | -0.1 (2.5) | -0.2 (2.0) | 0.2 (2.3) | 0.8 (2.4) | 0.1 (2.2)
  Chloride SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Chloride SFU | 1.0 (1.6) | 3.0 (2.7) | 0.5 (5.4) | 2.0 (0.0) | 0.0 (NA) — Value was not evaluable because only one participant was analyzed. | 0.3 (2.1)
  Potassium Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Potassium Week 1 | 0.08 (0.45) | 0.08 (0.33) | 0.05 (0.41) | 0.02 (0.36) | -0.03 (0.32) | 0.04 (0.29)
  Potassium Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Potassium Week 2 | 0.03 (0.30) | 0.08 (0.33) | 0.02 (0.32) | -0.06 (0.29) | 0.05 (0.37) | -0.03 (0.39)
  Potassium Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Potassium Week 4 | 0.09 (0.40) | 0.12 (0.41) | 0.09 (0.38) | 0.01 (0.34) | 0.05 (0.40) | 0.03 (0.33)
  Potassium Week 6: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Potassium Week 6 | -0.04 (0.32) | 0.11 (0.35) | -0.03 (0.31) | -0.07 (0.33) | -0.07 (0.34) | -0.02 (0.35)
  Potassium Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Potassium Week 8 | 0.01 (0.39) | 0.07 (0.36) | 0.12 (0.38) | -0.06 (0.38) | -0.12 (0.40) | 0.02 (0.35)
  Potassium Week 12: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 39
  Potassium Week 12 | -0.05 (0.35) | 0.08 (0.34) | 0.08 (0.37) | -0.06 (0.37) | -0.07 (0.37) | -0.06 (0.33)
  Potassium SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Potassium SFU | 0.10 (0.36) | 0.10 (0.37) | -0.10 (0.29) | -0.45 (0.07) | 0.20 (NA) — Value was not evaluable because only one participant was analyzed. | -0.20 (0.30)
  Magnesium Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Magnesium Week 1 | -0.010 (0.074) | -0.002 (0.052) | -0.020 (0.069) | 0.005 (0.079) | -0.007 (0.077) | -0.009 (0.064)
  Magnesium Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 42 | 42
  Magnesium Week 2 | -0.012 (0.063) | -0.004 (0.064) | -0.010 (0.065) | 0.001 (0.068) | -0.017 (0.086) | 0.005 (0.075)
  Magnesium Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Magnesium Week 4 | -0.023 (0.077) | -0.004 (0.062) | -0.017 (0.046) | 0.008 (0.071) | -0.017 (0.067) | -0.013 (0.070)
  Magnesium Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Magnesium Week 6 | -0.013 (0.054) | -0.014 (0.053) | -0.013 (0.057) | -0.008 (0.065) | -0.020 (0.073) | -0.017 (0.063)
  Magnesium Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Magnesium Week 8 | -0.026 (0.070) | -0.023 (0.042) | -0.023 (0.063) | 0.003 (0.071) | -0.019 (0.072) | -0.021 (0.058)
  Magnesium Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Magnesium Week 12 | -0.014 (0.093) | 0.007 (0.074) | -0.025 (0.069) | 0.009 (0.074) | -0.017 (0.075) | -0.008 (0.056)
  Magnesium SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Magnesium SFU | 0.053 (0.093) | 0.110 (0.295) | -0.035 (0.047) | -0.050 (0.057) | -0.060 (NA) — Value was not evaluable because only one participant was analyzed. | -0.023 (0.025)
  Sodium Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Sodium Week 1 | -0.1 (1.8) | 0.2 (1.7) | 0.3 (2.7) | 0.1 (1.9) | 0.0 (2.2) | 0.0 (1.4)
  Sodium Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 42 | 42
  Sodium Week 2 | -0.3 (1.7) | -0.2 (1.4) | -0.4 (1.8) | 0.0 (2.0) | 0.2 (2.3) | 0.0 (1.5)
  Sodium Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Sodium Week 4 | -0.2 (1.7) | 0.2 (1.7) | 0.2 (1.7) | -0.2 (1.7) | -0.1 (2.3) | -0.2 (1.7)
  Sodium Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Sodium Week 6 | -0.5 (2.0) | -0.1 (2.1) | -0.8 (1.6) | -0.1 (1.9) | -0.1 (2.9) | -0.3 (1.7)
  Sodium Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Sodium Week 8 | -0.6 (2.0) | 0.0 (2.8) | -0.2 (1.8) | -0.2 (2.0) | -0.1 (2.2) | -0.6 (2.0)
  Sodium Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Sodium Week 12 | -0.4 (2.0) | -0.2 (1.7) | -0.1 (1.7) | -0.2 (2.0) | -0.2 (2.4) | -0.3 (1.9)
  Sodium SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Sodium SFU | -0.5 (2.1) | 0.8 (1.7) | -2.0 (2.2) | -2.0 (2.8) | -1.0 (NA) — Value was not evaluable because only one participant was analyzed. | -1.7 (1.2)
  Urea Nitrogen Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Urea Nitrogen Week 1 | -0.16 (1.09) | 0.11 (1.12) | 0.27 (1.19) | 0.34 (1.22) | 0.27 (1.24) | 0.21 (0.88)
  Urea Nitrogen Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Urea Nitrogen Week 2 | 0.00 (1.16) | -0.03 (1.25) | 0.24 (1.16) | 0.16 (1.17) | 0.27 (1.17) | 0.37 (1.03)
  Urea Nitrogen Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Urea Nitrogen Week 4 | -0.14 (1.16) | 0.48 (1.52) | 0.50 (1.31) | -0.03 (1.20) | -0.11 (1.08) | 0.15 (1.04)
  Urea Nitrogen Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Urea Nitrogen Week 6 | -0.12 (0.96) | 0.21 (1.40) | 0.41 (1.14) | 0.19 (1.31) | 0.29 (1.14) | 0.12 (0.93)
  Urea Nitrogen Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Urea Nitrogen Week 8 | -0.28 (1.29) | 0.14 (1.33) | 0.32 (1.08) | -0.08 (1.58) | 0.33 (1.30) | 0.35 (0.88)
  Urea Nitrogen Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Urea Nitrogen Week 12 | -0.17 (1.35) | -0.04 (1.37) | 0.39 (1.14) | 0.08 (1.13) | 0.13 (1.08) | 0.01 (0.85)
  Urea Nitrogen SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Urea Nitrogen SFU | 0.65 (1.74) | 0.80 (1.19) | 0.78 (3.27) | -0.65 (2.05) | -0.30 (NA) — Value was not evaluable because only one participant was analyzed. | 0.77 (1.27)
  Cholesterol Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Cholesterol Week 1 | -0.04 (0.47) | -0.06 (0.54) | 0.00 (0.65) | -0.09 (0.59) | 0.12 (0.65) | 0.06 (0.34)
  Cholesterol Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Cholesterol Week 2 | -0.13 (0.71) | 0.03 (0.63) | 0.12 (0.58) | -0.11 (0.52) | 0.12 (1.04) | 0.05 (0.57)
  Cholesterol Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Cholesterol Week 4 | -0.06 (0.59) | 0.04 (0.63) | 0.17 (0.55) | -0.31 (0.88) | 0.00 (1.30) | 0.05 (0.66)
  Cholesterol Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Cholesterol Week 6 | 0.05 (0.46) | -0.02 (0.73) | 0.17 (0.56) | -0.24 (0.70) | -0.24 (1.32) | 0.08 (0.60)
  Cholesterol Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Cholesterol Week 8 | -0.08 (0.67) | -0.17 (0.68) | 0.16 (0.64) | -0.13 (0.83) | -0.17 (1.22) | 0.01 (0.48)
  Cholesterol Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Cholesterol Week 12 | -0.20 (0.88) | -0.07 (0.62) | 0.11 (0.62) | -0.18 (0.77) | 0.01 (1.29) | -0.05 (0.76)
  Cholesterol SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Cholesterol SFU | -0.28 (0.30) | -0.83 (1.56) | 0.38 (0.52) | -0.80 (0.14) | 0.20 (NA) — Value was not evaluable because only one participant was analyzed. | 0.40 (0.44)
  Glucose Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 42
  Glucose Week 1 | 0.50 (1.59) | 0.12 (0.82) | -0.14 (1.00) | -0.06 (1.14) | 0.07 (1.10) | 0.22 (0.70)
  Glucose Week 2: number analyzed (Participants) | 41 | 39 | 41 | 39 | 42 | 42
  Glucose Week 2 | 0.29 (1.62) | 0.17 (1.23) | -0.05 (0.92) | -0.20 (1.13) | 0.03 (1.09) | 0.05 (0.67)
  Glucose Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Glucose Week 4 | 0.37 (1.42) | 0.25 (1.22) | -0.12 (1.03) | -0.09 (1.24) | 0.37 (1.20) | 0.19 (0.92)
  Glucose Week 6: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Glucose Week 6 | 0.44 (1.42) | 0.30 (1.15) | -0.04 (1.26) | 0.02 (1.60) | 0.21 (1.30) | 0.29 (1.27)
  Glucose Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Glucose Week 8 | 0.37 (1.48) | 0.22 (1.48) | -0.15 (0.87) | -0.06 (1.43) | 0.11 (1.10) | 0.03 (0.97)
  Glucose Week 12: number analyzed (Participants) | 39 | 37 | 38 | 35 | 40 | 39
  Glucose Week 12 | 0.22 (1.27) | 0.01 (1.08) | 0.02 (1.35) | -0.17 (1.23) | -0.15 (0.88) | 0.04 (0.95)
  Glucose SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Glucose SFU | -0.40 (0.48) | 0.75 (0.89) | -0.33 (0.67) | -0.25 (0.49) | 0.20 (NA) — Value was not evaluable because only one participant was analyzed. | -0.17 (0.61)

23. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Lactate Dehydrogenase, Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Gamma Glutamyl Transferase)
Description: Lactate dehydrogenase, alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase and gamma glutamyl transferase were measured in units per liter (U/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
U/L
  Lactate Dehydrogenase Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Lactate Dehydrogenase Week 1 | -2.0 (29.4) | 1.1 (24.8) | -5.0 (24.1) | -0.3 (21.4) | -4.6 (18.9) | -3.4 (19.7)
  Lactate Dehydrogenase Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Lactate Dehydrogenase Week 2 | -4.9 (26.4) | -2.5 (25.2) | -3.5 (22.1) | 0.4 (27.6) | -7.6 (27.4) | -5.1 (20.1)
  Lactate Dehydrogenase Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Lactate Dehydrogenase Week 4 | -4.9 (22.4) | 1.7 (31.9) | -8.1 (16.7) | 5.0 (43.5) | -4.5 (37.7) | -4.4 (15.4)
  Lactate Dehydrogenase Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Lactate Dehydrogenase Week 6 | -5.0 (27.7) | -1.4 (25.2) | -7.3 (20.3) | 2.0 (16.2) | -11.0 (27.5) | -3.5 (22.6)
  Lactate Dehydrogenase Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Lactate Dehydrogenase Week 8 | -5.5 (27.4) | 0.5 (25.2) | -12.3 (22.2) | -0.8 (18.9) | -10.7 (33.1) | -3.7 (27.5)
  Lactate Dehydrogenase Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Lactate Dehydrogenase Week 12 | -4.9 (28.1) | 2.9 (26.7) | -7.5 (25.1) | -0.3 (20.6) | -5.6 (33.1) | -4.4 (24.8)
  Lactate Dehydrogenase SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Lactate Dehydrogenase SFU | -1.5 (12.9) | -5.0 (18.4) | 3.3 (81.2) | -45.5 (16.3) | 15.0 (NA) — Value was not evaluable because only one participant was analyzed. | 32.3 (34.2)
  Alkaline Phosphatase Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Alkaline Phosphatase Week 1 | -1.8 (6.3) | -0.5 (6.0) | -3.5 (8.2) | -3.8 (7.7) | -1.9 (5.3) | -2.3 (5.7)
  Alkaline Phosphatase Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Alkaline Phosphatase Week 2 | -3.0 (12.7) | 0.0 (7.4) | -2.5 (10.5) | -2.7 (8.2) | -1.6 (6.5) | -1.7 (7.7)
  Alkaline Phosphatase Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Alkaline Phosphatase Week 4 | -2.4 (8.7) | -1.9 (9.2) | -6.2 (9.8) | -4.3 (9.4) | -2.6 (8.1) | -1.7 (7.8)
  Alkaline Phosphatase Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Alkaline Phosphatase Week 6 | -3.0 (8.3) | -1.8 (9.0) | -5.5 (10.0) | -2.4 (8.6) | -2.1 (9.6) | -1.4 (7.5)
  Alkaline Phosphatase Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Alkaline Phosphatase Week 8 | -4.3 (12.2) | -1.7 (8.0) | -4.2 (11.2) | -2.1 (10.0) | -1.1 (11.3) | -1.9 (7.2)
  Alkaline Phosphatase Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Alkaline Phosphatase Week 12 | -2.0 (8.1) | 0.3 (7.2) | -2.4 (11.8) | -0.4 (9.0) | -0.5 (10.4) | -0.4 (8.4)
  Alkaline Phosphatase SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Alkaline Phosphatase SFU | -0.5 (7.4) | 9.8 (8.9) | 7.8 (15.3) | -3.0 (5.7) | 3.0 (NA) — Value was not evaluable because only one participant was analyzed. | 3.0 (1.0)
  Alanine Aminotransferase Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Alanine Aminotransferase Week 1 | 2.0 (7.7) | 2.1 (10.4) | -1.7 (13.7) | 1.6 (12.2) | 0.7 (8.9) | 1.2 (9.1)
  Alanine Aminotransferase Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Alanine Aminotransferase Week 2 | 0.3 (6.5) | 1.9 (9.0) | 2.0 (29.8) | -0.9 (7.7) | -0.2 (10.2) | 1.6 (11.5)
  Alanine Aminotransferase Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Alanine Aminotransferase Week 4 | -0.2 (7.0) | 1.1 (8.6) | 0.8 (18.7) | -0.4 (10.2) | 0.4 (14.7) | 1.0 (13.3)
  Alanine Aminotransferase Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Alanine Aminotransferase Week 6 | 3.9 (18.9) | 1.1 (8.9) | -0.6 (11.7) | 3.5 (20.9) | -1.7 (13.7) | 1.1 (12.5)
  Alanine Aminotransferase Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Alanine Aminotransferase Week 8 | 1.8 (10.8) | 2.2 (10.2) | 0.1 (10.5) | -0.4 (9.7) | -1.1 (14.5) | 0.8 (9.0)
  Alanine Aminotransferase Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Alanine Aminotransferase Week 12 | -1.3 (7.5) | 1.8 (9.9) | -1.0 (10.8) | -0.9 (9.1) | -0.9 (14.6) | -0.4 (10.6)
  Alanine Aminotransferase SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Alanine Aminotransferase SFU | -3.8 (3.0) | 4.3 (3.4) | 26.5 (42.1) | -6.0 (8.5) | 16.0 (NA) — Value was not evaluable because only one participant was analyzed. | -3.3 (3.1)
  Aspartate Aminotransferase Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Aspartate Aminotransferase Week 1 | 0.5 (6.1) | 2.0 (10.8) | -3.0 (15.2) | 1.9 (11.5) | 0.3 (6.3) | -0.5 (7.2)
  Aspartate Aminotransferase Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Aspartate Aminotransferase Week 2 | -1.0 (3.8) | 0.4 (4.9) | -1.9 (19.1) | -0.9 (4.7) | -0.5 (6.1) | 0.9 (13.4)
  Aspartate Aminotransferase Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Aspartate Aminotransferase Week 4 | -1.1 (4.8) | -0.1 (5.8) | -2.5 (17.5) | -0.4 (5.9) | 0.6 (8.2) | -0.4 (7.5)
  Aspartate Aminotransferase Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Aspartate Aminotransferase Week 6 | 1.5 (10.6) | 0.8 (6.0) | -0.9 (9.5) | 4.0 (15.7) | -1.4 (7.0) | -1.4 (6.5)
  Aspartate Aminotransferase Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Aspartate Aminotransferase Week 8 | 0.0 (5.1) | 0.2 (6.7) | -1.4 (5.4) | -1.4 (4.6) | -0.4 (8.3) | -0.8 (6.3)
  Aspartate Aminotransferase Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Aspartate Aminotransferase Week 12 | -1.3 (5.5) | 1.1 (7.9) | -1.4 (8.3) | -0.3 (4.8) | -0.5 (7.3) | -0.9 (5.2)
  Aspartate Aminotransferase SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Aspartate Aminotransferase SFU | -2.8 (1.7) | -0.3 (2.1) | 11.5 (23.5) | -4.0 (2.8) | 9.0 (NA) — Value was not evaluable because only one participant was analyzed. | 0.7 (2.5)
  Gamma Glutamyl Transferase Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Gamma Glutamyl Transferase Week 1 | 0.6 (6.4) | -0.8 (14.1) | -2.0 (10.7) | -7.5 (42.1) | 1.6 (22.9) | -0.8 (6.3)
  Gamma Glutamyl Transferase Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Gamma Glutamyl Transferase Week 2 | 0.2 (8.7) | -1.6 (11.1) | 0.2 (14.2) | -1.2 (8.0) | -1.9 (6.5) | 0.4 (15.0)
  Gamma Glutamyl Transferase Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Gamma Glutamyl Transferase Week 4 | -0.7 (8.5) | -1.9 (11.8) | 1.8 (18.6) | -2.6 (12.8) | -0.4 (8.4) | -1.4 (14.1)
  Gamma Glutamyl Transferase Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Gamma Glutamyl Transferase Week 6 | 1.8 (10.5) | -1.8 (13.8) | -2.9 (13.1) | -2.9 (7.3) | -2.1 (9.3) | -1.1 (12.9)
  Gamma Glutamyl Transferase Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Gamma Glutamyl Transferase Week 8 | 2.4 (13.7) | -1.9 (14.9) | -0.9 (18.4) | -2.6 (13.6) | -2.5 (9.4) | 3.1 (29.5)
  Gamma Glutamyl Transferase Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Gamma Glutamyl Transferase Week 12 | -0.4 (10.9) | -2.2 (13.3) | -1.1 (21.7) | -0.6 (11.2) | -0.4 (11.1) | -0.9 (12.2)
  Gamma Glutamyl Transferase SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Gamma Glutamyl Transferase SFU | -8.0 (13.4) | 1.3 (3.9) | 19.8 (23.3) | -16.5 (24.7) | 37.0 (NA) — Value was not evaluable because only one participant was analyzed. | 3.0 (3.5)

24. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (Creatinine, Bilirubin)
Description: Creatinine and bilirubin were measured in micromols per liter (μmol/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
μmol/L
  Creatinine Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Creatinine Week 1 | 0.6 (7.0) | 2.7 (10.1) | 1.4 (8.6) | 0.6 (8.1) | 0.7 (8.4) | -0.7 (7.7)
  Creatinine Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Creatinine Week 2 | 0.0 (7.1) | -0.8 (8.2) | -0.4 (10.1) | -0.7 (8.5) | -0.1 (8.3) | 0.0 (7.1)
  Creatinine Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Creatinine Week 4 | 0.0 (5.8) | 1.3 (9.1) | 0.6 (7.9) | -1.7 (8.1) | 0.6 (8.1) | 1.6 (7.2)
  Creatinine Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Creatinine Week 6 | -1.1 (7.8) | 1.6 (10.5) | -0.1 (10.6) | -0.6 (7.9) | -0.1 (8.1) | -0.5 (11.1)
  Creatinine Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Creatinine Week 8 | -1.1 (6.2) | -0.4 (7.4) | -1.0 (9.6) | -2.6 (8.4) | -0.1 (7.6) | 0.1 (8.3)
  Creatinine Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Creatinine Week 12 | -1.6 (7.8) | -0.2 (7.0) | 0.7 (12.0) | -0.7 (9.1) | 0.1 (9.0) | -0.7 (7.2)
  Creatinine SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Creatinine SFU | 1.5 (4.4) | 6.0 (4.3) | -6.5 (4.4) | -10.5 (16.3) | 9.0 (NA) — Value was not evaluable because only one participant was analyzed. | 1.3 (6.4)
  Bilirubin Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Bilirubin Week 1 | -0.53 (3.10) | -1.79 (4.50) | -0.52 (2.81) | -0.55 (4.49) | 0.57 (5.73) | 0.14 (4.16)
  Bilirubin Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Bilirubin Week 2 | -0.35 (2.85) | -0.86 (5.05) | -0.48 (3.40) | -0.38 (3.60) | -0.99 (2.98) | 0.27 (3.69)
  Bilirubin Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 41
  Bilirubin Week 4 | -0.70 (3.26) | -1.70 (4.92) | -0.26 (3.53) | -0.04 (2.74) | 0.76 (4.27) | 0.70 (4.52)
  Bilirubin Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Bilirubin Week 6 | -0.51 (3.13) | -1.15 (4.59) | 0.35 (3.44) | -0.33 (3.94) | 0.11 (4.19) | -0.30 (4.28)
  Bilirubin Week 8: number analyzed (Participants) | 39 | 38 | 38 | 34 | 40 | 40
  Bilirubin Week 8 | -0.21 (3.81) | -0.98 (4.68) | -0.30 (3.20) | -0.43 (4.52) | -0.15 (3.79) | -0.02 (4.41)
  Bilirubin Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Bilirubin Week 12 | -0.74 (3.43) | -1.02 (5.24) | -0.73 (2.98) | -1.20 (3.37) | -0.43 (3.68) | -0.34 (3.45)
  Bilirubin SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Bilirubin SFU | 2.05 (2.16) | -1.23 (2.62) | -0.30 (3.87) | -0.25 (0.78) | -1.50 (NA) — Value was not evaluable because only one participant was analyzed. | 1.40 (2.96)

25. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Biochemistry Parameters (C Reactive Protein)
Description: C Reactive Protein was measured in milligrams per liters (mg/L).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
mg/L
  Week 1: number analyzed (Participants) | 15 | 10 | 6 | 8 | 12 | 10
  Week 1 | -2.110 (5.255) | -5.367 (11.806) | -0.775 (2.020) | -2.635 (2.550) | -5.108 (10.013) | -3.732 (3.997)
  Week 2: number analyzed (Participants) | 11 | 10 | 7 | 9 | 9 | 9
  Week 2 | 1.821 (6.974) | -6.985 (11.064) | 0.576 (2.898) | 2.743 (15.212) | -6.763 (13.211) | -3.042 (1.989)
  Week 4: number analyzed (Participants) | 11 | 10 | 6 | 7 | 10 | 8
  Week 4 | 1.338 (11.182) | -5.835 (8.594) | -1.722 (5.596) | 0.929 (8.047) | -4.226 (9.865) | 7.141 (32.344)
  Week 6: number analyzed (Participants) | 14 | 8 | 7 | 4 | 8 | 6
  Week 6 | 2.978 (13.162) | -5.930 (9.560) | -4.516 (11.304) | -0.595 (7.346) | 1.799 (14.635) | -6.598 (6.278)
  Week 8: number analyzed (Participants) | 12 | 8 | 7 | 4 | 9 | 5
  Week 8 | 3.153 (18.764) | -6.891 (15.192) | -3.143 (10.844) | 2.590 (7.755) | 12.434 (47.447) | -1.104 (5.201)
  Week 12: number analyzed (Participants) | 10 | 11 | 6 | 4 | 8 | 8
  Week 12 | 7.279 (13.546) | -5.193 (10.817) | 0.695 (6.381) | -3.033 (7.261) | -9.890 (10.729) | -5.368 (5.322)
  SFU: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
  SFU | 8.000 (NA) — Value was not evaluable because only one participant was analyzed. |  |  |  |  |

26. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Urinalysis Parameters (pH)
Description: Urine pH was measured on a pH scale.
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: ph
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
ph
  Week 1: number analyzed (Participants) | 42 | 39 | 41 | 40 | 43 | 43
  Week 1 | 0.00 (0.79) | -0.10 (0.79) | -0.13 (0.88) | -0.20 (0.88) | -0.08 (0.82) | -0.07 (0.90)
  Week 2: number analyzed (Participants) | 42 | 39 | 39 | 39 | 42 | 42
  Week 2 | 0.06 (0.86) | -0.06 (0.86) | -0.10 (0.77) | -0.23 (0.92) | -0.18 (0.76) | 0.06 (0.65)
  Week 4: number analyzed (Participants) | 41 | 39 | 41 | 39 | 41 | 40
  Week 4 | 0.05 (0.87) | -0.09 (0.76) | -0.11 (0.95) | -0.26 (0.89) | -0.07 (0.73) | -0.04 (0.74)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | -0.01 (0.73) | -0.03 (0.68) | -0.17 (0.69) | -0.18 (0.86) | -0.13 (0.81) | 0.05 (0.86)
  Week 8: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 40
  Week 8 | -0.03 (0.92) | -0.07 (0.83) | -0.12 (1.07) | -0.34 (0.79) | -0.30 (0.91) | 0.08 (0.75)
  Week 12: number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
  Week 12 | -0.14 (0.79) | -0.01 (0.85) | 0.01 (0.70) | -0.28 (0.85) | -0.21 (0.99) | -0.01 (0.85)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 0.25 (1.04) | -0.25 (0.87) | 0.50 (1.22) | -1.00 (1.41) | 0.50 (NA) — Value was not evaluable because only one participant was analyzed. | -0.17 (0.29)

27. Secondary Outcome: Percentage of Participants Who Shifted From Baseline Until Week 12 in Urinalysis Parameters (Leukocyte Esterase)
Description: Percentages were based on the number of participants with non-missing urinalysis results at Baseline and at Week 12.
Time Frame: From Baseline (Week 0) until Week 12
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
  Number of participants reflect those with non-missing urinalysis results at Baseline and at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
percentage of participants
  Baseline Low - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 High | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Normal | 84.6 | 84.2 | 97.3 | 88.2 | 90.0 | 92.3
  Baseline Normal - Week 12 High | 2.6 | 0 | 2.7 | 5.9 | 5.0 | 0
  Baseline High - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline High - Week 12 Normal | 7.7 | 15.8 | 0 | 2.9 | 5.0 | 7.7
  Baseline High - Week 12 High | 5.1 | 0 | 0 | 2.9 | 0 | 0

28. Secondary Outcome: Percentage of Participants Who Shifted From Baseline Until Week 12 in Urinalysis Parameters (Nitrite)
Description: Percentages were based on the number of participants with non-missing urinalysis results at Baseline and at Week 12.
Time Frame: From Baseline (Week 0) until Week 12
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
percentage of participants
  Baseline Low - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 High | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Normal | 97.4 | 97.4 | 100 | 100 | 95.0 | 94.9
  Baseline Normal - Week 12 High | 0 | 2.6 | 0 | 0 | 2.5 | 2.6
  Baseline High - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline High - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 2.6
  Baseline High - Week 12 High | 2.6 | 0 | 0 | 0 | 2.5 | 0

29. Secondary Outcome: Percentage of Participants Who Shifted From Baseline Until Week 12 in Urinalysis Parameters (Occult Blood)
Description: Percentages were based on the number of participants with non-missing urinalysis results at Baseline and at Week 12.
Time Frame: From Baseline (Week 0) until Week 12
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
percentage of participants
  Baseline Low - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 High | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Normal | 76.9 | 86.8 | 83.8 | 79.4 | 77.5 | 89.7
  Baseline Normal - Week 12 High | 0 | 5.3 | 0 | 5.9 | 5.0 | 2.6
  Baseline High - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline High - Week 12 Normal | 10.3 | 5.3 | 5.4 | 8.8 | 15.0 | 5.1
  Baseline High - Week 12 High | 12.8 | 2.6 | 10.8 | 5.9 | 2.5 | 2.6

30. Secondary Outcome: Percentage of Participants Who Shifted From Baseline Until Week 12 in Urinalysis Parameters (Urine Glucose)
Description: Percentages were based on the number of participants with non-missing urinalysis results at Baseline and at Week 12.
Time Frame: From Baseline (Week 0) until Week 12
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
percentage of participants
  Baseline Low - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 High | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Normal | 94.9 | 94.7 | 97.3 | 97.1 | 95.0 | 94.9
  Baseline Normal - Week 12 High | 0 | 2.6 | 2.7 | 2.9 | 0 | 0
  Baseline High - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline High - Week 12 Normal | 0 | 0 | 0 | 0 | 2.5 | 0
  Baseline High - Week 12 High | 5.1 | 2.6 | 0 | 0 | 2.5 | 5.1

31. Secondary Outcome: Percentage of Participants Who Shifted From Baseline Until Week 12 in Urinalysis Parameters (Albumin)
Description: Percentages were based on the number of participants with non-missing urinalysis results at Baseline and at Week 12.
Time Frame: From Baseline (Week 0) until Week 12
Population: as for outcome 27
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 39 | 38 | 37 | 34 | 40 | 39
percentage of participants
  Baseline Low - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 Normal | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Low - Week 12 High | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline Normal - Week 12 Normal | 94.9 | 89.5 | 86.5 | 91.2 | 95.0 | 92.3
  Baseline Normal - Week 12 High | 0 | 7.9 | 2.7 | 2.9 | 2.5 | 0
  Baseline High - Week 12 Low | 0 | 0 | 0 | 0 | 0 | 0
  Baseline High - Week 12 Normal | 5.1 | 2.6 | 10.8 | 5.9 | 2.5 | 2.6
  Baseline High - Week 12 High | 0 | 0 | 0 | 0 | 0 | 5.1

32. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Vital Signs (Blood Pressure)
Description: Blood pressure was measured in millimeters of mercury (mmHg).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
mmHg
  Systolic Blood Pressure Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Systolic Blood Pressure Week 1 | 1.2 (10.7) | 2.2 (7.1) | -3.9 (8.3) | 1.7 (9.3) | 0.2 (12.1) | -1.0 (9.9)
  Systolic Blood Pressure Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Systolic Blood Pressure Week 2 | -1.1 (9.7) | 2.1 (9.4) | -2.7 (12.5) | 0.2 (13.6) | -0.6 (8.4) | -3.2 (11.2)
  Systolic Blood Pressure Week 4: number analyzed (Participants) | 42 | 39 | 41 | 39 | 41 | 41
  Systolic Blood Pressure Week 4 | -2.3 (10.0) | 2.1 (7.9) | -1.9 (11.3) | 0.1 (12.4) | -0.1 (11.3) | -0.5 (10.8)
  Systolic Blood Pressure Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Systolic Blood Pressure Week 6 | -1.4 (9.8) | -1.3 (10.7) | -4.3 (10.6) | 0.1 (12.8) | -0.9 (10.9) | -2.4 (9.2)
  Systolic Blood Pressure Week 8: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Systolic Blood Pressure Week 8 | -0.8 (12.1) | -1.3 (13.0) | -3.4 (8.0) | 0.1 (12.3) | 0.5 (12.5) | -1.0 (10.7)
  Systolic Blood Pressure Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Systolic Blood Pressure Week 12 | -1.3 (10.9) | 2.2 (9.0) | -2.9 (10.3) | -0.3 (11.8) | -1.2 (10.4) | -2.4 (10.1)
  Systolic Blood Pressure SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Systolic Blood Pressure SFU | -7.0 (12.7) | -10.5 (17.0) | -1.3 (10.4) | 4.5 (7.8) | -2.0 (NA) — Value was not evaluable because only one participant was analyzed. | -2.0 (2.6)
  Diastolic Blood Pressure Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Diastolic Blood Pressure Week 1 | -0.4 (7.4) | 0.9 (10.0) | -2.1 (7.3) | 0.6 (6.5) | 0.3 (7.4) | 0.1 (6.7)
  Diastolic Blood Pressure Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Diastolic Blood Pressure Week 2 | -1.5 (6.9) | 0.4 (8.7) | -1.2 (7.1) | 2.1 (8.3) | 0.0 (7.2) | 0.2 (7.0)
  Diastolic Blood Pressure Week 4: number analyzed (Participants) | 42 | 39 | 41 | 39 | 41 | 41
  Diastolic Blood Pressure Week 4 | -0.3 (7.8) | 0.6 (9.2) | -0.3 (7.9) | 0.6 (7.3) | 0.0 (7.7) | 0.3 (8.1)
  Diastolic Blood Pressure Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Diastolic Blood Pressure Week 6 | 0.3 (7.6) | 0.0 (9.7) | -3.1 (7.9) | 1.3 (8.6) | 0.1 (7.3) | -1.6 (7.3)
  Diastolic Blood Pressure Week 8: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Diastolic Blood Pressure Week 8 | -1.1 (8.9) | -0.3 (9.1) | -1.2 (7.3) | 2.8 (8.7) | -0.7 (7.7) | -0.6 (8.2)
  Diastolic Blood Pressure Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Diastolic Blood Pressure Week 12 | -2.3 (5.8) | 0.5 (6.3) | -1.7 (6.4) | 3.1 (8.4) | -1.1 (6.7) | -1.1 (7.3)
  Diastolic Blood Pressure SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  Diastolic Blood Pressure SFU | 1.3 (8.5) | -9.0 (9.1) | 0.8 (8.8) | -4.5 (0.7) | -9.0 (NA) — Value was not evaluable because only one participant was analyzed. | -4.0 (6.6)

33. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Vital Signs (Pulse Rate)
Description: Pulse rate was measured in beats per minute (beats/min).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
beats/min
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Week 1 | 1.7 (9.5) | -1.6 (9.1) | 3.2 (8.0) | -1.8 (8.1) | 0.1 (6.4) | -0.4 (7.7)
  Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Week 2 | 1.2 (8.4) | -1.3 (9.9) | 1.1 (7.8) | -1.0 (10.4) | -2.2 (7.9) | 0.5 (9.5)
  Week 4: number analyzed (Participants) | 42 | 39 | 41 | 39 | 41 | 41
  Week 4 | 1.0 (10.2) | -3.1 (9.9) | 0.6 (7.8) | -3.6 (9.0) | -1.6 (6.5) | 1.6 (8.0)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | 0.9 (9.8) | 1.2 (10.7) | 1.4 (8.3) | -2.6 (9.7) | -1.7 (9.3) | 2.6 (8.0)
  Week 8: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Week 8 | 1.7 (8.9) | -3.2 (9.3) | 0.4 (9.2) | -1.8 (8.5) | 0.5 (8.2) | 0.6 (6.7)
  Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Week 12 | 0.9 (8.4) | -1.9 (6.8) | 1.8 (11.0) | -3.1 (8.5) | -1.7 (9.1) | 0.0 (7.5)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | -2.8 (2.6) | -2.5 (12.0) | 2.3 (6.0) | 1.5 (4.9) | -7.0 (NA) — Value was not evaluable because only one participant was analyzed. | 7.3 (3.2)

34. Secondary Outcome: Change From Baseline Until Safety Follow-up Visit in Vital Signs (Temperature)
Description: Temperature was measured in degrees Celsius (°C).
Time Frame: as for outcome 15
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
°C
  Week 1: number analyzed (Participants) | 42 | 39 | 42 | 40 | 43 | 43
  Week 1 | -0.07 (0.23) | -0.04 (0.22) | 0.02 (0.30) | -0.11 (0.32) | -0.07 (0.30) | 0.02 (0.35)
  Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Week 2 | 0.00 (0.26) | 0.02 (0.26) | 0.01 (0.33) | 0.01 (0.35) | -0.04 (0.36) | -0.01 (0.35)
  Week 4: number analyzed (Participants) | 42 | 39 | 41 | 39 | 41 | 41
  Week 4 | -0.05 (0.29) | 0.03 (0.24) | 0.00 (0.42) | -0.04 (0.24) | -0.03 (0.26) | -0.01 (0.41)
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 37 | 40 | 40
  Week 6 | -0.03 (0.29) | -0.02 (0.25) | -0.01 (0.22) | -0.06 (0.43) | -0.03 (0.38) | 0.07 (0.24)
  Week 8: number analyzed (Participants) | 39 | 38 | 38 | 37 | 40 | 40
  Week 8 | 0.01 (0.24) | -0.02 (0.28) | 0.00 (0.33) | -0.03 (0.41) | 0.00 (0.35) | 0.02 (0.31)
  Week 12: number analyzed (Participants) | 39 | 38 | 38 | 35 | 40 | 39
  Week 12 | 0.10 (0.27) | 0.00 (0.27) | 0.06 (0.36) | -0.04 (0.28) | 0.00 (0.33) | 0.00 (0.30)
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 0.08 (0.22) | 0.15 (0.33) | -0.03 (0.05) | 0.10 (0.00) | 0.10 (NA) — Value was not evaluable because only one participant was analyzed. | 0.43 (0.31)

35. Secondary Outcome: Percentage of Participants With Clinically Significant Physical Examination Abnormalities
Description: The physical examination included general appearance; ear, nose, and throat; eyes, hair, and skin; respiratory; CV; GI; musculoskeletal; hepatic; neurological (including limb reflexes); and mental status.
  Any clinically significant abnormal findings during the study were captured as adverse events.
Time Frame: At Screening, Week 12/Early Withdrawal Visit and the Safety Follow-Up Visit (20 weeks after the last dose)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants | 23.8 | 7.7 | 11.6 | 10.0 | 9.3 | 0

36. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: Percentages were based on the number of participants with a non-missing measurement for that variable at the visit.
Time Frame: Baseline (Week 0), Week 2, Week 4, Week 6, Week 12, and Safety Follow-Up visit (20 weeks after the last dose)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 160 mg w/ LD Q4W (SS) | Bimekizumab 320 mg Q4W (SS) | Bimekizumab 480 mg Q4W (SS)
Number analyzed (Participants) | 42 | 39 | 43 | 40 | 43 | 43
percentage of participants
  Baseline | 0 | 0 | 0 | 2.5 | 0 | 0
  Week 2: number analyzed (Participants) | 42 | 39 | 41 | 39 | 42 | 42
  Week 2 | 0 | 0 | 0 | 2.6 | 0 | 0
  Week 4: number analyzed (Participants) | 42 | 39 | 41 | 39 | 41 | 41
  Week 4 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 40 | 38 | 38 | 36 | 40 | 40
  Week 6 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 39 | 38 | 38 | 34 | 39 | 39
  Week 12 | 0 | 0 | 0 | 0 | 0 | 0
  SFU: number analyzed (Participants) | 4 | 4 | 4 | 2 | 1 | 3
  SFU | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from Baseline (Week 0) to End of Safety Follow-up (up to Week 28)
Description: It was pre-specified to report adverse events (AE) that have a start date on or following the first administration of study treatment. TEAEs counts are for each study period: Treatment Period (Wk1-12) for all participants who received at least 1 study treatment and Post-Treatment Period for participants who either enrolled in an extension study (PS0011) or those who entered a 20-week Safety Follow-Up Period.
Groups:
- Placebo (SS) Treatment Period: During the Treatment Period participants randomized to the placebo group, received a combination of several injections of placebo, subcutaneously every 4 weeks (Q4W). Participants formed the Safety Set (SS).
- Bimekizumab 64 mg Q4W (SS) Treatment Period: During the Treatment Period participants were randomized to receive subcutaneous injections of 64 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 160 mg Q4W (SS) Treatment Period: During the Treatment Period participants were randomized to receive subcutaneous injections of 160 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 160 mg w/ LD Q4W (SS) Treatment Period: During the Treatment Period participants were randomized to receive subcutaneous injections of 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 320 mg Q4W (SS) Treatment Period: During the Treatment Period participants were randomized to receive subcutaneous injections of 320 mg bimekizumab Q4W. Participants formed the SS.
- Bimekizumab 480 mg Q4W (SS) Treatment Period: During the Treatment Period participants were randomized to receive subcutaneous injections of 480 mg bimekizumab Q4W. Participants formed the SS.
- Placebo (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive Placebo during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
- Bimekizumab 64 mg Q4W (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive 64 mg bimekizumab Q4W during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
- Bimekizumab 160 mg Q4W (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive 160 mg bimekizumab Q4W during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
- Bimekizumab 160 mg w/ LD Q4W (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive 320 mg bimekizumab loading dose at Baseline followed by 160 mg bimekizumab Q4W during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
- Bimekizumab 320 mg Q4W (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive 320 mg bimekizumab Q4W during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
- Bimekizumab 480 mg Q4W (SS) Post-Treatment Period: At Week 12, participants who were randomized to receive 480 mg bimekizumab Q4W during the Treatment Period and who enrolled in the extension study (PS0011), underwent the Week 12 study assessments and then received their first extension study dose of study treatment. All participants who did not enroll in the extension study had the Week 12 study assessments and entered the Safety Follow-Up (SFU) Period, 20 weeks after the last dose of study medication.
  Participants did not receive any treatment during the Post-Treatment Period. Participants formed the SS.
Arm/Group | Placebo (SS) Treatment Period | Bimekizumab 64 mg Q4W (SS) Treatment Period | Bimekizumab 160 mg Q4W (SS) Treatment Period | Bimekizumab 160 mg w/ LD Q4W (SS) Treatment Period | Bimekizumab 320 mg Q4W (SS) Treatment Period | Bimekizumab 480 mg Q4W (SS) Treatment Period | Placebo (SS) Post-Treatment Period | Bimekizumab 64 mg Q4W (SS) Post-Treatment Period | Bimekizumab 160 mg Q4W (SS) Post-Treatment Period | Bimekizumab 160 mg w/ LD Q4W (SS) Post-Treatment Period | Bimekizumab 320 mg Q4W (SS) Post-Treatment Period | Bimekizumab 480 mg Q4W (SS) Post-Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39 | 0/43 | 0/40 | 0/43 | 0/43 | 0/42 | 0/39 | 0/43 | 0/40 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/39 | 0/43 | 0/40 | 0/43 | 1/43 | 0/42 | 1/39 | 0/43 | 0/40 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 8/42 | 16/39 | 12/43 | 12/40 | 14/43 | 10/43 | 0/42 | 0/39 | 0/43 | 0/40 | 0/43 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) Treatment Period (N=42) | Bimekizumab 64 mg Q4W (SS) Treatment Period (N=39) | Bimekizumab 160 mg Q4W (SS) Treatment Period (N=43) | Bimekizumab 160 mg w/ LD Q4W (SS) Treatment Period (N=40) | Bimekizumab 320 mg Q4W (SS) Treatment Period (N=43) | Bimekizumab 480 mg Q4W (SS) Treatment Period (N=43) | Placebo (SS) Post-Treatment Period (N=42) | Bimekizumab 64 mg Q4W (SS) Post-Treatment Period (N=39) | Bimekizumab 160 mg Q4W (SS) Post-Treatment Period (N=43) | Bimekizumab 160 mg w/ LD Q4W (SS) Post-Treatment Period (N=40) | Bimekizumab 320 mg Q4W (SS) Post-Treatment Period (N=43) | Bimekizumab 480 mg Q4W (SS) Post-Treatment Period (N=43)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) Treatment Period (N=42) | Bimekizumab 64 mg Q4W (SS) Treatment Period (N=39) | Bimekizumab 160 mg Q4W (SS) Treatment Period (N=43) | Bimekizumab 160 mg w/ LD Q4W (SS) Treatment Period (N=40) | Bimekizumab 320 mg Q4W (SS) Treatment Period (N=43) | Bimekizumab 480 mg Q4W (SS) Treatment Period (N=43) | Placebo (SS) Post-Treatment Period (N=42) | Bimekizumab 64 mg Q4W (SS) Post-Treatment Period (N=39) | Bimekizumab 160 mg Q4W (SS) Post-Treatment Period (N=43) | Bimekizumab 160 mg w/ LD Q4W (SS) Post-Treatment Period (N=40) | Bimekizumab 320 mg Q4W (SS) Post-Treatment Period (N=43) | Bimekizumab 480 mg Q4W (SS) Post-Treatment Period (N=43)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (5) | 3 (3) | 3 (3) | 6 (6) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 2 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT02905006/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT02905006/SAP_001.pdf